CLINICAL TRIAL: NCT06889961
Title: Effect of Daily Mixed Spice Consumption on Memory in Middle-Aged and Older Adults with Age-related Cognitive Decline: a Pilot Study
Brief Title: Effect of Daily Mixed Spice Consumption on Memory Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine and Chief of the Division of Clinical Nutrition at the University of California, Los Angeles, University of California, Los Angeles
Allocation: Not Applicable | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 23-001878
Record Dates: First submitted 2025-02-25; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Memory; Cognitive Function

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mixed spices (Active Comparator)
  Interventions: Dietary Supplement: Mixed spices
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Mixed spices — Mixed spices 4.00 g capsules of spice mixture contain 1.0 g (25%) turmeric, 1.5 g (37.5%) cinnamon, 0.5 g (12.5%) oregano, 0.5 g (12.5%) black pepper, 0.3 g (7.5%) sage and 0.2 (5%) thyme
  Arms: Mixed spices
Other: Placebo — 4.00 g maltodextrin capsules
  Arms: Placebo

SUMMARY:
The aging process entails a multitude of structural and functional alterations within the brain, culminating in a gradual and progressive decline in cognitive function. Recent research has indicated that various spices may hold the key to enhancing brain health and combating the effects of aging on cognitive abilities. The hypothesis is that a mixture of spices, acknowledged for their reported memory protection potential, may yield a more potent beneficial effect on memory function than a single spice. The spice mixture will be used at culinary dose, and therefore side effects are anticipated. In this study, the effects of spice mixture will be evaluated, as well as their anti-oxidant, and anti-inflammatory properties. The proposed pilot study will include 50 adults (ages 50-80), exhibiting typical age-related mild cognitive decline, excluding dementia or major neurocognitive disorders. They will be randomized 1:1 assigned into a daily intake of either 4.00 g spice mixture capsules or 4.00 g maltodextrin capsules over 3 months, and explore the sustainable effect over 3 additional months. The changes in symptoms of cognition, fatigue, and mood symptoms of the spice group vs. placebo group will be compared. The outcome of the investigation of the effects of mixed spice consumption will provide important novel information on dietary recommendation of spice to preserve cognitive function in aging population.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are required to have clinical histories consistent with normal aging or mild cognitive impairment (MCI).
2. Age 50 to 80 years.
3. Adequate visual acuity and hearing to allow neuropsychological testing.
4. Screening laboratory tests without significant abnormalities that might interfere with the study.

   -

Exclusion Criteria:

1. Diagnosis of probable Alzheimer's disease or any other dementia (e.g. vascular, Lewy body, frontotemporal)
2. Evidence of other neurological or physical illness that can produce cognitive deterioration. Determination of dementia will be based on the clinical evaluation including assessment of functional abilities, and cognitive screening (using the Mini Mental State Examination
3. Evidence of Parkinson's disease as determined by the motor examination (items 18-31) of the Unified Parkinson's Disease Rating Scale [38].
4. Uncontrolled hypertension (systolic blood pressure (BP) > 170 or diastolic BP > 100).
5. Consume spices regularly > 5g day
6. Allergy or sensitivity to spices. Subjects will be excluded if there is a prior history of such sensitivity. Since these foods are commonly eaten and allergies are rare, subjects should be aware of this sensitivity prior to entering the study. To determine this, a positive history of spices ingestion without incident will be requested. In addition, any subject with a history of allergy or anaphylaxis of any kind will be excluded.
7. Current diagnosis of any major psychiatric disorder according to the DSM-IV TR criteria (APA, 2000).
8. Current diagnosis or alcoholism or substance addiction.
9. Eating a high fiber/polyphenol diet or taking any medication or dietary supplement which interfere with the absorption of polyphenols.
10. Frequently using prebiotics, probiotics, yogurt, and/or any fiber supplements

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2027-02-21 (Estimated); Study Completion 2027-02-21 (Estimated)

PRIMARY OUTCOMES:
Memory | 6 month
  Verbal Episodic Memory (Rey Auditory Verbal Learning Test (RAVLT)-Revised, number of words correctly recalled after the long delay).

SECONDARY OUTCOMES:
Executive Function | 6 month
  These will be measured by Trailmaking part B (time/seconds) and Wechsler Adult Intelligence Scale Version IV (WAIS-IV), DVT (Digit Span Backwards). The length of the battery is approximately 15 minutes.
Language, Executive Function, Episodic Memory, Processing Speed, and Working Memory | 6 month
  Language, Executive Function, Episodic Memory, Processing Speed, and Working Memory will also be evaluated by The NIH Toolbox Cognition Battery (NIHTB-CB) It can be administered via computer, paper and pencil, and most recently, ipad platforms (45 mins). We will analyze, as a secondary outcome measure, the Crystallized Intelligence index.
Fatigue | 6 month
  Fatigue (as assessed by PROMIS-Fatigue Scale, Short Form 8 items): The NIH developed Patient Reported Outcomes Measurement Information System (PROMIS®). The PROMIS Fatigue scale assess a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. The fatigue short forms are universal rather than disease-specific and assess fatigue over the past seven days (5 minutes).
Body weight | 6 month
  Body weight: Body weight will be measured at baseline, 6,12, and 24 weeks.
Body composition | 6 month
  Body composition: Body weight and composition analysis will be performed using the Tanita-BC418 body-fat analyzer (Tanita Corp., Tokyo, Japan) based on the principles of bioelectrical impedance at baseline, 6,12, and 24 weeks.
Sleep Quality | 6 month
  Sleep Quality, Pittsburgh Sleep Quality Index: PSQI will be employed to assess sleep quality. The PSQI is a widely recognized self-report questionnaire that evaluates sleep quality over a one-month interval. The PSQI comprises 19 self-rated items and an additional 5 items rated by bed partners or roommates. The self-rated items are used to calculate the total score, which ranges from 0 to 21. Each item on the PSQI is scored on a scale of 0 to 3, with 3 reflecting the highest level of dysfunction or disturbance. The scores of these items are then summed to compute a global PSQI score. A global PSQI score greater than 5 suggests significant sleep difficulties. A higher total score is indicative of poorer sleep quality.
24-hour Diet Recall | 6 month
  24-hour Diet Recall: Dietary energy and macronutrient intake will be assessed at baseline, 6,12, and 24 weeks during site visits. For the 24-hr dietary recall we will be using the Automated Self-Administered 24-hour Dietary Recall (ASA24™) tool (https://asa24.nci.nih.gov/).
Quality of life, SF-36 | 6 month
  The SF-36 domain:
  Physical Functioning: Measures the ability to perform a range of physical activities without limitations, such as walking, climbing stairs, or carrying groceries.
Quality of life, SF-36 | 6 month
  The SF-36 domain:
  Role-Physical: Assesses limitations in work or daily activities due to physical health problems.
Quality of life, SF-36 | 6 month
  The SF-36 domain:
  Pain: Evaluates the impact of pain on daily activities and the extent of pain experienced.
Quality of life, SF-36 | 6 month
  The SF-36 domain:
  General Health: Reflects overall health perceptions, including personal health outlook and resistance to illness.
Quality of life, SF-36 | 6 month
  The SF-36 domain:
  Vitality: Captures energy levels and fatigue, distinguishing between feeling energetic versus feeling tired or worn out.
Quality of life, SF-36 | 6 month
  The SF-36 domain:
  Social Functioning: Measures the impact of physical or emotional health on social activities and interactions with others.
Quality of life, SF-36 | 6 month
  The SF-36 domain:
  Role-Emotional: Assesses the extent to which emotional problems interfere with work or other daily activities.
Quality of life, SF-36 | 6 month
  The SF-36 domain:
  Mental Health: Evaluates psychological well-being, including feelings of depression, anxiety, and overall emotional stability.

OTHER OUTCOMES:
Blood anti-oxidation capacity | 6 month
  Blood anti-oxidation capacity will be measured using Oxygen radical antioxidant capacity (ORAC) and trolox equivalent antioxidant capacity (TEAC) assays.
Plasma inflammatory panel | 6 month
  Plasma inflammatory panel will be measured using the Luminex MagPix® analyzer (Luminex, Austin TX)
Fecal microbiome | 6 month
  Fecal microbiome will be analyzed at UCLA microbiome core
Mitochondrial function | 6 month
  Mitochondrial function as well as aging markers will be evaluated using blood samples at the UCLA Mitochondrial Metabolism core and Center for Human Nutrition Analytical Laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutrition, Los Angeles, California, United States